CLINICAL TRIAL: NCT02472158
Title: Use of Chlorhexidine-gel-Impregnated Dressing Compared to Transparent Polyurethane Film Dressing as Coverage of the Site of Insertion of Central Venous Catheter, in the Evaluation of Catheter Colonization in Critically Ill Adults Patients: A Randomized Controlled Trial
Brief Title: Chlorhexidine-Impregnated Sponge Dressing: A Clinical Trial
Acronym: CISDCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Amanda Salles Margatho, PhD Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CISD-15
Record Dates: First submitted 2015-01-26; First posted 2015-06-15 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Catheter-Related Infections
Keywords: Bandages; Central Venous Catheters; Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- chlorhexidine-gel-impregnated dressing (Experimental): Chlorhexidine Patients receive a chlorhexidine-gel-impregnated dressing ( 3M Tegaderm CHG IV securement dressing™ ) after insertion of central venous catheter
  Interventions: Device: chlorhexidine-gel-impregnated dressing
- Polyurethane film dressing (Active Comparator): Polyurethane film dressing Patients receive a transparent polyurethane film dressing (3M Tegaderm IV dressing™) after insertion of central venous catheter.
  Interventions: Device: Polyurethane film dressing

INTERVENTIONS:
Device: chlorhexidine-gel-impregnated dressing — Chlorhexidine Patients receive a chlorhexidine-gel-impregnated dressing ( 3M Tegaderm CHG IV securement dressing™ ) after insertion of central venous catheter
  Other Names: 3M Tegaderm CHG IV securement dressing™
  Arms: chlorhexidine-gel-impregnated dressing
Device: Polyurethane film dressing — Polyurethane film dressing Patients receive a transparent polyurethane film dressing (3M Tegaderm IV dressing™) after insertion of central venous catheter.
  Other Names: 3M Tegaderm IV dressing™
  Arms: Polyurethane film dressing

SUMMARY:
The purpose of this study is to compare the use of chlorhexidine-gel-impregnated dressing and the transparent polyurethane film dressing as coverage of the site of insertion of central venous catheter, in the evaluation of catheter colonization in critically ill adults patients.

ELIGIBILITY:
Inclusion Criteria:

Critically ill patients hospitalized carrying a short-term central venous catheter

Exclusion Criteria:

* Use of a central venous catheter with antimicrobial coating
* Suspected or confirmed bacterial infection at randomization
* Known allergic/hypersensitivity reaction to any compounds of the treatment
* Active lesions in the skin where the CVC is located and / or where the dressing of CVC is being conducted;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Catheter Colonization | Participants will be followed from placement until the withdraw of the central venous catheter, an expected average of 3 weeks.
  With aseptic technique, the central venous catheter will be withdrawn and a 5 centimeters distal portion of the catheter will be cut and conditioned in sterile test tube and sent to the microbiology laboratory. It will be considered a Catheter Colonization a significant growth of one or more microorganism in a semiquantitative culture of the catheter tip. It is according to the Clinical Practice Guidelines for the Diagnosis and management of Intravascular Catheter- Related Infection: 2009 Update by the Infectious Diseases Society of America

SECONDARY OUTCOMES:
Microbiological Exit site Infection | Participants will be followed from placement until the withdraw of central venous catheter, an expected average of 3 weeks
  With aseptic technique, a swab will be collected before removal of central venous catheter, the swab will be moistened with sterile saline and rolled for about 2 cm around the exit site. The material will be conditioned in sterile test tube and sent to the microbiology laboratory. It will be considered a Microbiological Exit Site Infection the exudate at catheter exit site yields a microorganism. According to Clinical Practice Guideline for Diagnosis and Management of intravascular Catheter-Related Infection: 2009 Update by the Infectious Diseases Society of America
Clinical Exit Site Infection | Participants will be followed from placement until the withdraw of central venous catheter, an expected average of 3 weeks
  Erythema, induration, and/or tenderness within 2 cm of the catheter exit site, according to Clinical Practice Guidelines for the diagnosis and management of intravascular Catheter-Related Infection: 2009 Update by the infectious diseases Society of America.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Salles Margatho, PhD student, Study Chair — University of São Paulo at Ribeirão Preto College of Nursing
Locations (1):
- Clinical Hospital of Ribeirão Preto Medical School (HCFMRP-USP), Ribeirão Preto, São Paulo, Brazil